CLINICAL TRIAL: NCT04273997
Title: Randomised, Double-blind, Placebo-controlled Trial Evaluating the Effects of Metronidazole Ointment in Facilitating Resolution of Non-healing Pilonidal Sinus Wounds.
Brief Title: Metronidazole Ointment in Non-healing Pilonidal Sinus Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: S.L.A. Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MET-PS-02
Record Dates: First submitted 2020-01-15; First posted 2020-02-18 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus | interventions — Metronidazole; Ointments

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled trial evaluating the effects of metronidazole ointment in facilitating resolution of non-healing pilonidal sinus wounds
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole Ointment (Active Comparator): Treatment Group A: Metronidazole 10% w/w ointment. A 2.5 cm strip of ointment (approximately 700 mg) will be administered topically to the wound together with suitable dressing, once daily.
  One dose contains approximately 70 mg metronidazole in a formulation of white soft paraffin. The Investigator will demonstrate to the subject how to apply a 2.5 cm of IMP and dress the wound by applying the first dose and covering with a dry, gauze dressing which is to be retained with tape. Larger wounds may require additional amount of IMP to ensure sufficient cover of the wound
  Interventions: Drug: Metronidazole 10% ointment
- Placebo Ointment (Placebo Comparator): Treatment Group B: Placebo ointment. A 2.5 cm strip of ointment (approximately 700 mg) will be administered topically to the wound together with suitable dressing, once daily.
  One dose of placebo ointment contains titanium dioxide and white soft paraffin. The Investigator will demonstrate to the subject how to apply a 2.5 cm of IMP and dress the wound by applying the first dose and covering with a dry, gauze dressing which is to be retained with tape. Larger wounds may require additional amount of IMP to ensure sufficient cover of the wound.
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Metronidazole 10% ointment — Metronidazole 10% ointment
  Other Names: Ortem
  Arms: Metronidazole Ointment
Drug: Placebo ointment — Placebo ointment
  Arms: Placebo Ointment

SUMMARY:
Title of Study:

Randomised, double-blind, placebo-controlled trial evaluating the effects of metronidazole ointment in facilitating resolution on non-healing pilonidal sinus wounds Medical Condition Under Investigation Non-healing pilonidal sinus wounds

Study centres: 2 Centres in Turkey

Clinical Phase: Phase 2

Protocol Number: MET-PS-02

Study Design: Randomised, double-blind, placebo-controlled, parallel group study to determine the safety and efficacy of metronidazole ointment applied to the wound, following debridement in non-healing pilonidal sinus wounds.

Planned Sample Size: 80 subjects

DETAILED DESCRIPTION:
Route of Administration: Cutaneous

Investigational product and dosage:

Treatment Group A: Metronidazole 10% w/w ointment. A 2.5 cm strip of ointment (approximately 700 mg) will be administered topically to the wound together with suitable dressing, once daily.

One dose contains approximately 70 mg metronidazole in a formulation of white soft paraffin. The Investigator will demonstrate to the subject how to apply a 2.5 cm of IMP and dress the wound by applying the first dose and covering with a dry, gauze dressing which is to be retained with tape. Larger wounds may require additional amount of IMP to ensure sufficient cover of the wound.

Comparator and dosage:

Treatment Group B: Placebo ointment. A 2.5 cm strip of ointment (approximately 700 mg) will be administered topically to the wound together with suitable dressing, once daily.

One dose of placebo ointment contains titanium dioxide and white soft paraffin. The Investigator will demonstrate to the subject how to apply a 2.5 cm of IMP and dress the wound by applying the first dose and covering with a dry, gauze dressing which is to be retained with tape. Larger wounds may require additional amount of IMP to ensure sufficient cover of the wound.

Maximum Duration of Treatment:

The subject's participation in the study will last 10 weeks (including 2 week screening, 6 weeks clinical phase and 2 week follow-up phase).

Procedures:

Recruitment:

Subjects will be recruited through surgical out-patient clinics who will be contacted directly or through advertisements. Potential Subjects will have the opportunity to read or hear the study advertisement and contact the researcher through the contact details provided. Potential participants will have the opportunity to ask any questions to the researchers.

A member of the research team will then send a copy of the information sheet (either by email or post) or hand to the participant, who will have the opportunity to ask any questions to the researchers, either by email or phone.

Subjects expressing an interest in participating will be interviewed at their scheduled clinic appointment to explain the study in detail, and discuss the risks, benefits, goals and limitations of the study by the treating nurse.

Screening:

Potentially eligible Subjects will provide written informed consent prior to any study specific procedures being conducted.

Following the provision of written, informed consent, the Subject's demography, medical history, especially that relating to pilonidal sinus including details on surgical interventions, will be documented. Female Subjects of child-bearing potential will undergo a urine pregnancy test. Following a physical examination, height, weight and checks on vital signs, the Subjects will have blood samples drawn for routine haematology and biochemistry analyses. Subjects will be asked to provide details of any concomitant medications. The wound will be sized and graded using the Pressure Ulcer Scale for Healing (PUSH) tool 3.0. Subjects will have their wound assessed, then debrided and any surrounding hair removed by shaving, cleaned and dressed in accordance with normal management procedures.

Subjects with a confirmed diagnosis of non-healing pilonidal sinus wound, compliance with the inclusion and exclusion criteria and providing written informed consent will be registered on the electronic case report form (eCRF) to obtain a screening number.

The Investigator will demonstrate to the subject how to clean and dress the wound.

The subject will be educated on the use of the diary and asked to record at the end of each day the number of times they cleaned and dressed the wound and any changes in their condition or concomitant medication. Subjects will be asked to complete the diary over the subsequent 2 weeks.

Subjects not wishing to participate, or who are ineligible, will be followed up in accordance with the clinic's standard management procedures.

Baseline:

The subject will attend the clinic and the diary will be reviewed to ensure completion of the diary, the number of times the wound was cleaned and dressed, any changes in their condition or concomitant medications. Haematology and biochemistry test (from Screening) results will be confirmed as being acceptable.

Subjects will have the status of their pilonidal disease assessed and the wound will be sized and graded using the Pressure Ulcer Scale for Healing (PUSH) tool 3.0, to confirm that it remains unhealed with no improvement.

Subjects demonstrating improvement in the wound and healing in the screening period, will be followed up in accordance with the clinic's standard management procedures.

Female Subjects of child-bearing potential will undergo a pregnancy test. Subjects compliant with the inclusion and exclusion criteria will be randomised on a 1:1 basis to one of the two treatment groups: metronidazole 10%w/w ointment or matching placebo ointment. Randomisation will be stratified by wound size less than 3cm.

Following a physical examination, weight and checks on vital signs, blood samples will be drawn for routine haematology and biochemistry analyses. The wound will be swabbed for microbial analysis, then debrided and any surrounding hair removed by shaving.

The subject will be provided with two pre-weighed tubes of IMP together with a supply of sterile dressings. The Investigator will demonstrate to the subject how to apply 2.5 cm of IMP and dress the wound by applying the first dose and covering with a dry, gauze dressing which is to be retained with tape.

The subject will be retrained on completion of the diary and asked to record each day confirmation of wound cleansing, IMP dose application and wound dressing as well as any changes in their condition or concomitant medication.

Week 1:

One week after randomisation, the subject will be contacted by telephone to check on their progress, compliance with study medication, concomitant medications and the occurrence of any adverse events.

Weeks 2, 4 and 6 :

Two, four and six weeks after randomisation, the subject will attend the clinic for review of the healing status of their pilonidal disease including sizing of the wound and assignment of a PUSH score, together with checks on vital signs and a physical examination. In addition, the subject will complete the PGI I in relation to their pilonidal disease, relative to the baseline condition.

Haematology and biochemistry test (from Baseline) results will be confirmed as being acceptable (Week 2 Visit only).

At each visit the IMP tubes will be weighed to determine the amount used as a check on compliance with study treatment. The subject diary will be reviewed and any changes in symptoms and concomitant medications registered in the eCRF.

The Investigator will clean the wound and remove any surrounding hair by shaving. During each visit apply the dose of IMP and dress the wound for that day (Week 2 and Week 4 Visits only).

At the Week 6 visit, subjects will also provide blood samples for routine haematology and biochemistry analyses. Female subjects of child-bearing potential will undergo a pregnancy test. Subjects considered a clinical failure will have the pilonidal sinus wound swabbed for microbiological analysis.

In the event that the wound is judged to be completely healed at any visit, the subject will be instructed to stop applying the study medication. The Week 6 procedures will be performed and the subject will be asked to attend the clinic after a further 2 weeks, when the Week 8 procedures will be undertaken.

In the event that a subject wishes to withdraw prior to the end of the study, they will be asked to undertake the Week 6 procedures.

For subjects who have failed to heal, appropriate post-study treatment will be instituted.

Week 8 (follow-up):

Eight weeks after randomisation (or two weeks after a visit at which complete healing is confirmed), the subject will attend the clinic for review of the healing status of the pilonidal disease including wound size and PUSH score, together with checks on vital signs, changes in symptoms and concomitant medications. The subject will complete the PGI I in relation to their pilonidal disease, relative to the baseline condition. Haematology and biochemistry test (from Week 6 Visit) results will be confirmed as being acceptable.

Blood and urine sampling:

A blood sample will be drawn at the Screening, Baseline and Week 6 Visits for routine haematology and biochemistry tests.

Urine pregnancy tests will be conducted at Screening, Baseline and Week 6 Visits.

Safety Parameters:

Study subjects will be asked to record any changes in symptoms in the diary provided on a daily basis. This will be reviewed at each study visit and any adverse events will be documented in the eCRF. Changes in vital signs and outcome of routine blood analyses will be evaluated.

Adverse events (AEs) will be classified using a coding thesaurus (MedDRA).

Primary Endpoint:

Complete wound healing by Week 6.

Secondary Endpoints:

* Rate of wound healing [(baseline mm3 - Current mm3) / baseline mm3 x 100%
* Proportion of subjects with complete healing by Week 2 and 4
* Proportion of subjects with complete healing maintained over two consecutive visits
* Time to response, defined as complete healing
* Change from baseline in PUSH score at Weeks 2, 4 and 6
* Patient's Global Impression of Improvement (PGI-I) at Weeks 2, 4 and 6

Safety Endpoints:

The safety analysis will be conducted in all randomised subjects receiving at least one dose.

* Number and proportion of subjects with adverse events.
* Assessment of clinical laboratory parameters.
* Assessment of vital signs.

Statistical Analyses:

Proportion of subjects with complete healing and with partial healing will be presented using point estimates with 95% confidence intervals.

Differences in the rates of healing will be determined by difference in the mean. SE of the mean and 95% confidence interval will be reported.

Time to response will be presented in Kaplan-Meier curves. PUSH score will be presented by using point estimates with 95% confidence intervals. Comparisons between each treatment and placebo will be based on an Analysis of covariance (ANCOVA) model.

PGI-I will be presented by category using point estimates with 95% confidence intervals. Comparisons between each treatment and placebo will be based on a proportional odds model.

AEs will be classified into standard terminology using a coding thesaurus (MedDRA). Treatment-related AEs will be summarised separately from all AEs. In addition, the maximum intensity of AEs will be summarised. For AEs these will be summarized using descriptive statistics. Results of laboratory tests and measures of vital signs will be presented as summary statistics and as shift tables.

Missing data will be handled using a worst observation carried forward (WOCF) imputation. Sensitivity analyses will be included in the SAP.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent.
2. Male or female aged ≥18 years.
3. Previous surgery for pilonidal disease and failure of healing for ≥ 6 weeks post-surgical excision of the pilonidal cyst/sinus;
4. Willingness to stop all other concomitant topical preparations at the site of pilonidal sinus wounds.

Exclusion criteria:

The subject will be excluded from the study if any of the following applies:

1. Presence of non-drained abscess (abscess must have been drained ≥ 6 weeks prior to entry).
2. Subjects who are due to undergo surgery related to pilonidal sinus.
3. Previous use (in the last 2 weeks) or current treatment with any antibiotic. To be determined by medical history prior to screening.
4. Previous treatment with topical metronidazole for pilonidal sinus.
5. Known allergic reaction to metronidazole.
6. Known allergic reaction to excipients of IMP and placebo.
7. Subject is taking any prohibited medication (warfarin-type anticoagulants, fluorouracil, glucocorticoids, other topical preparations to the area of the wound, lithium, cyclosporin and disulfiram).
8. Experimental agents must have been discontinued at least 8 weeks prior to screening or for a period equivalent to 5 half-lives of the agent (whichever is longer).
9. History of epilepsy or seizures.
10. Subject has hepatic insufficiency as defined by laboratory values outside the normal ranges.
11. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless surgically sterile must use effective contraception (either combined oestrogen and progestogen containing hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD], intrauterine hormone-releasing system [IUS], vasectomised partner, sexual abstinence (only considered an acceptable method of contraception when it is in line with the subjects' usual and preferred lifestyle), combination of male condom with either cap, diaphragm or sponge with spermicide [double barrier methods]), and willing and able to continue contraception for 1 month after the last administration of IMP. Women using oral contraception must have started using it at least 2 months prior to screening. Women are not considered to be of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels that have been confirmed to be in the "postmenopausal range". Or have had a surgical bilateral oophorectomy (with or without hysterectomy) or bilateral tubal ligation at least six weeks before the screening visit. In case of oophorectomy alone, the reproductive status of the woman should have been confirmed by follow up hormone level assessment.
12. Women who are pregnant or breastfeeding at baseline.
13. Subjects with concurrent disease considered by the Investigator to be clinically significant in the context of the study.
14. Subjects who have clinically significant abnormalities on their screening blood tests. "Clinically significant" will be determined by the surgeon at the study site.
15. Subjects who will be unavailable for the duration of the trial, deemed unable to comply with the requirements of the study protocol, likely to be noncompliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason.
16. Subjects who show a 20% reduction in wound size between screening and baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete healing by Week 6. | 6 weeks
  Proportion of subjects treated with Metronidazole ointment to placebo with complete healing by Week 6.

SECONDARY OUTCOMES:
Determine the effects of Metronidazole ointment on the time course of healing • Determine the effects of metronidazole in promoting partial healing | 2-6 weeks
  Rate of wound healing [(baseline mm3 - Current mm3) / baseline mm3 x 100%
Subjects with complete healing by weeks 2 and 4 | 2-4 weeks
  Proportion of subjects with complete healing by Week 2 and 4
Maintaining of complete healing over consecutive visits | 2-6 weeks
  Proportion of subjects with complete healing maintained over two consecutive visits
response time for complete healing | 2-6 weeks
  Time to response, defined as complete healing
PUSH score change | weeks 2, 4 and 6
  Change from baseline in PUSH score at Weeks 2, 4 and 6
Determine the effects of metronidazole on the patient's global impression of improvement | weeks 2, 4 and 6
  Patient's Global Impression of Improvement (PGI-I) at Weeks 2, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Arda Isik, Principal Investigator — Study Principal Investigator; Ozan Kucuk, Principal Investigator — Study Principal Investigator
Locations (2):
- Turkey (Türkiye) (2):
  - Erzincan Binali Yıldırım University General Surgery Clinic, Erzincan
  - Samsun Training and Research Hospital General Surgery Clinic, Samsun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akinci OF, Bozer M, Uzunkoy A, Duzgun SA, Coskun A. Incidence and aetiological factors in pilonidal sinus among Turkish soldiers. Eur J Surg. 1999 Apr;165(4):339-42. doi: 10.1080/110241599750006875. PMID 10365835
- [Background] Ala S, Saeedi M, Eshghi F, Mirzabeygi P. Topical metronidazole can reduce pain after surgery and pain on defecation in postoperative hemorrhoidectomy. Dis Colon Rectum. 2008 Feb;51(2):235-8. doi: 10.1007/s10350-007-9174-3. Epub 2008 Jan 4. PMID 18176825
- [Background] Maeda Y, Ng SC, Durdey P, Burt C, Torkington J, Rao PK, Mayberry J, Moshkovska T, Stone CD, Carapeti E, Vaizey CJ; Topical Metronidazole in Perianal Crohn's Study Group. Randomized clinical trial of metronidazole ointment versus placebo in perianal Crohn's disease. Br J Surg. 2010 Sep;97(9):1340-7. doi: 10.1002/bjs.7121. PMID 20632322
- [Background] Saidy M, Ali A, Adewole A, Ambroze W, Schertzer M, King E, Armstrong D. (2016) Treatment of non-healing pilonidal disease using topical 10% metronidazole: a 10-year review. Annual scientific meeting American Society Colon and Rectal surgeon (ASCRS), April 30-May 4, Los Angeles, USA.
- [Background] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Background] Ypsilantis E, Carapeti E, Chan S. The use of topical 10% metronidazole in the treatment of non-healing pilonidal sinus wounds after surgery. Int J Colorectal Dis. 2016 Mar;31(3):765-7. doi: 10.1007/s00384-015-2269-8. Epub 2015 May 24. No abstract available. PMID 26003119